CLINICAL TRIAL: NCT03908476
Title: PROLONG Prospective, Multi-center, Open-label, Post-market Study
Acronym: PROLONG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ABT-CIP-10277
Record Dates: First submitted 2019-03-13; First posted 2019-04-09 (Actual); Results first posted 2023-01-25 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Chronic Pain
Keywords: Chronic Pain; Spinal cord stimulation; ABT-CIP-10277; BurstDR; SCS; DRG
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Subjects using BurstDR SCS systems (Experimental): Spinal cord stimulation with a Burst waveform.
  Interventions: Device: Burst-capable SCS system
- Subjects using DRG systems (Experimental): Dorsal root ganglion stimulation.
  Interventions: Device: DRG Stimulator

INTERVENTIONS:
Device: Burst-capable SCS system — Subjects will be given Burst stimulation using a market-released Abbott SCS system. Burst stimulation may be achieved through surgical or non-surgical means.
  Arms: Subjects using BurstDR SCS systems
Device: DRG Stimulator — Subjects will be implanted with a market-released Abbott DRG stimulation system.
  Arms: Subjects using DRG systems

SUMMARY:
Spinal cord stimulation (SCS) has been shown to be effective for relieving intractable chronic pain. However, a portion of patients who initially succeed with SCS will eventually lose their therapeutic benefit. Reliable methods have not been identified for restoring neuromodulation benefit to this underserved population, so additional research is required. This study will prospectively observe subjects who utilize Abbott neurostimulation devices after failing to sustain pain relief with their previous SCS system. The effectiveness of Abbott systems in restoring neuromodulation benefit will be evaluated over the course of a two-year follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must provide written informed consent prior to any clinical investigation related procedure.
2. Patient has a spinal cord stimulator implanted for chronic, intractable pain.
3. Patient has inadequate pain relief from their current SCS system.
4. Patient has a pain NRS ≥ 6.
5. Physician has determined that the patient's original pain is still addressable with neurostimulation.

Exclusion Criteria:

1. Patient is enrolled, or intends to participate, in a competing clinical study, as determined by Abbott.
2. Patient is seeking care for a new pain complaint outside of the original indication for SCS.
3. Presence of other anatomic or comorbid conditions, or other medical, social, or psychological conditions that, in the Investigator's opinion, could limit the patient's ability to participate in the clinical investigation or to comply with follow-up requirements.
4. Physician has determined that patient's pain relief is inadequate due to a malfunction or damage to the existing system.
5. Patient requires frequent MRI.
6. Patient is involved in active disability litigation related to their pain or seeking worker's compensation.
7. Patient is part of a vulnerable population.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2019-04-16 (Actual); Primary Completion 2021-11-15 (Actual); Study Completion 2021-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marie Fahey, Study Director — Abbott
Locations (21):
- United States (21):
  - Spanish Hills Interventional Pain Specialists, Camarillo, California
  - Coastal Pain & Spinal Diagnostics Medical Group, Carlsbad, California
  - UC San Diego Center for Pain Medicine, La Jolla, California
  - Napa Valley Orthopedic Medical Group, Napa, California
  - Newport Beach Headache & Pain, Newport Beach, California
  - Spine & Nerve Diagnostic Center, Roseville, California
  - Pacific Research Institute, San Francisco, California
  - Front Range Pain Medicine, Fort Collins, Colorado
  - Boca Raton Regional Hospital, Boca Raton, Florida
  - Pain Care, LLC, Stockbridge, Georgia
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Nura, Edina, Minnesota
  - Nevada Advanced Pain Specialists, Reno, Nevada
  - Garden State Pain Control, Clifton, New Jersey
  - Albany Medical College at Albany Medical Center, Albany, New York
  - Ainsworth Institute of Pain Management, New York, New York
  - Northwest Brain & Spine, Bend, Oregon
  - Center for Interventional Pain and Spine, Lancaster, Pennsylvania
  - Allegheny General Hospital Department of Neurosurgery, Pittsburgh, Pennsylvania
  - The Spine & Nerve Center of St. Francis Hospital, Charleston, West Virginia
  - St. Mary's Hospital, Huntington, West Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 100 subjects proceeded with a permanent implant
Period: Overall Study
Arm/Group | Subjects Using BurstDR SCS Systems | Subjects Using DRG Systems
Started | 85 | 15
Completed | 64 | 13
Not Completed | 21 | 2
Not completed — Death | 3 | 0
Not completed — Lost to Follow-up | 3 | 1
Not completed — Withdrawal by Subject | 7 | 1
Not completed — Physician Decision | 2 | 0
Not completed — System Explanted and not Replaced | 4 | 0
Not completed — Intrathecal Pump | 1 | 0
Not completed — Patient Has Requested an Explant of the Device | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Subjects Using BurstDR SCS Systems | Subjects Using DRG Systems | Total
Number analyzed (Participants) | 85 | 15 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.6 (12.8) | 57.2 (18.7) | 61.8 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 8 | 55
  Male | 38 | 7 | 45
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 76 | 12 | 88
  Unknown or Not Reported | 8 | 2 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 0 | 3
  White | 77 | 14 | 91
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 1 | 4
Region of Enrollment [Number; unit: participants]
  United States | 85 | 15 | 100

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Pain Assessed by Numerical Rating Scale (NRS) From Baseline to 3 Months
Description: Numerical Rating Scale (NRS) is a scale which measures pain intensity from 0-10, with 0 being no pain and 10 being worst pain.
Time Frame: From Baseline to 3 months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Subjects Using BurstDR SCS Systems | Subjects Using DRG Systems
Number analyzed (Participants) | 74 | 15
score on a scale | 2.3 (2.5) | 3.3 (2.7)

2. Primary Outcome: Mean Change in Pain Assessed by Numerical Rating Scale (NRS) From Baseline to 6 Months
Description: as for outcome 1
Time Frame: From Baseline to 6 months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Subjects Using BurstDR SCS Systems | Subjects Using DRG Systems
Number analyzed (Participants) | 67 | 14
score on a scale | 2.5 (2.7) | 3.1 (3.5)

3. Primary Outcome: Mean Change in Pain Assessed by Numerical Rating Scale (NRS) From Baseline to 12 Months
Description: as for outcome 1
Time Frame: From Baseline to 12 months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Subjects Using BurstDR SCS Systems | Subjects Using DRG Systems
Number analyzed (Participants) | 66 | 13
score on a scale | 2.5 (2.6) | 2.6 (3.3)

4. Primary Outcome: Mean Change in Pain Assessed by Numerical Rating Scale (NRS) From Baseline to 18 Months
Description: as for outcome 1
Time Frame: From Baseline to 18 months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Subjects Using BurstDR SCS Systems | Subjects Using DRG Systems
Number analyzed (Participants) | 45 | 11
score on a scale | 2.2 (2.5) | 1.5 (3.6)

5. Primary Outcome: Mean Change in Pain Assessed by Numerical Rating Scale (NRS) From Baseline to 24 Months
Description: as for outcome 1
Time Frame: From Baseline to 24 months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Subjects Using BurstDR SCS Systems | Subjects Using DRG Systems
Number analyzed (Participants) | 23 | 7
score on a scale | 2.8 (2.6) | 2.0 (2.4)

6. Secondary Outcome: Mean Change in Health Domains Assessed by PROMIS-29 Scale From Baseline to 3 Months
Description: Patient Reported Outcomes Measurement Information System Adult Profile The PROMIS-29 is a 29-item profile instrument that covers 7 health domains (depression, anxiety, physical function, pain interference, fatigue, sleep disturbance, and social function) with 4 questions each. The final item is an 11-point pain intensity numerical rating scale (NRS). Subjects should read each item and check the one box that most closely represents their response.
  Each item is scored on a scale from 1-5 with total scores for each domain ranging from 4-20. Greater scores represent more of whatever concept is being measured (e.g., depression or physical function). The scoring tables have been provided in the measure manual. Raw domain scores are converted to t-scores with a mean of 50 and a standard deviation of 10. The t-scores were validated on a sample from the general population and all items must be answered to utilize the scoring tables.
Time Frame: From baseline to 3 months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Subjects Using BurstDR SCS Systems | Subjects Using DRG Systems
Number analyzed (Participants) | 85 | 15
score on a scale
  Physical Function: number analyzed (Participants) | 74 | 15
  Physical Function | -2.72 (5.63) | -4.90 (7.93)
  Anxiety: number analyzed (Participants) | 74 | 15
  Anxiety | 2.36 (8.81) | 1.05 (7.18)
  Depression: number analyzed (Participants) | 73 | 15
  Depression | 3.02 (9.47) | 2.43 (9.12)
  Fatigue: number analyzed (Participants) | 74 | 15
  Fatigue | 3.03 (9.91) | 7.51 (6.87)
  Sleep Disturbance: number analyzed (Participants) | 74 | 15
  Sleep Disturbance | 4.08 (8.00) | 2.99 (10.91)
  Social Roles and Activities: number analyzed (Participants) | 74 | 15
  Social Roles and Activities | -3.25 (8.36) | -4.54 (11.52)
  Pain Interference: number analyzed (Participants) | 73 | 15
  Pain Interference | 5.00 (7.87) | 5.56 (9.25)
  Pain Intensity: number analyzed (Participants) | 74 | 15
  Pain Intensity | 1.9 (2.4) | 2.9 (2.3)

7. Secondary Outcome: Mean Change in Health Domains Assessed by PROMIS-29 Scale From Baseline to 6 Months
Description: as for outcome 6
Time Frame: From baseline to 6 months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Subjects Using BurstDR SCS Systems | Subjects Using DRG Systems
Number analyzed (Participants) | 85 | 15
score on a scale
  Physical Function: number analyzed (Participants) | 67 | 14
  Physical Function | -2.21 (5.28) | -5.30 (8.64)
  Anxiety: number analyzed (Participants) | 67 | 14
  Anxiety | 2.99 (7.64) | -0.96 (11.25)
  Depression: number analyzed (Participants) | 67 | 14
  Depression | 2.52 (8.74) | -1.78 (9.83)
  Fatigue: number analyzed (Participants) | 67 | 14
  Fatigue | 3.03 (9.55) | 4.81 (12.37)
  Sleep Disturbance: number analyzed (Participants) | 67 | 14
  Sleep Disturbance | 4.73 (9.59) | 4.23 (13.32)
  Social Roles and Activities: number analyzed (Participants) | 67 | 14
  Social Roles and Activities | -2.76 (8.04) | -4.49 (11.29)
  Pain Interference: number analyzed (Participants) | 67 | 14
  Pain Interference | 5.32 (7.44) | 6.59 (9.54)
  Pain Intensity: number analyzed (Participants) | 67 | 14
  Pain Intensity | 2.2 (2.4) | 3.0 (3.2)

8. Secondary Outcome: Mean Change in Health Domains Assessed by PROMIS-29 Scale From Baseline to 12 Months
Description: as for outcome 6
Time Frame: From baseline to 12 months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Subjects Using BurstDR SCS Systems | Subjects Using DRG Systems
Number analyzed (Participants) | 85 | 15
score on a scale
  Physical Function: number analyzed (Participants) | 66 | 13
  Physical Function | -2.28 (5.74) | -5.97 (8.01)
  Anxiety: number analyzed (Participants) | 66 | 13
  Anxiety | 1.96 (9.86) | 2.68 (12.71)
  Depression: number analyzed (Participants) | 66 | 13
  Depression | 1.05 (10.14) | 0.30 (11.43)
  Fatigue: number analyzed (Participants) | 66 | 13
  Fatigue | 3.38 (8.72) | 4.19 (10.76)
  Sleep Disturbance: number analyzed (Participants) | 66 | 13
  Sleep Disturbance | 3.44 (8.83) | 2.81 (12.24)
  Social Roles and Activities: number analyzed (Participants) | 66 | 13
  Social Roles and Activities | -2.13 (8.36) | -4.99 (11.01)
  Pain Interference: number analyzed (Participants) | 66 | 13
  Pain Interference | 4.68 (7.94) | 6.46 (11.16)
  Pain Intensity: number analyzed (Participants) | 66 | 13
  Pain Intensity | 2.0 (2.4) | 2.7 (3.1)

9. Secondary Outcome: Mean Change in Health Domains Assessed by PROMIS-29 Scale From Baseline to 18 Months
Description: as for outcome 6
Time Frame: From baseline to 18 months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Subjects Using BurstDR SCS Systems | Subjects Using DRG Systems
Number analyzed (Participants) | 85 | 15
score on a scale
  Physical Function: number analyzed (Participants) | 45 | 11
  Physical Function | -1.20 (5.37) | -4.02 (7.81)
  Anxiety: number analyzed (Participants) | 45 | 11
  Anxiety | 1.22 (10.94) | 3.04 (8.29)
  Depression: number analyzed (Participants) | 45 | 11
  Depression | 1.39 (9.64) | 1.04 (5.21)
  Fatigue: number analyzed (Participants) | 45 | 11
  Fatigue | 1.39 (9.51) | 6.04 (11.27)
  Sleep Disturbance: number analyzed (Participants) | 45 | 11
  Sleep Disturbance | 3.55 (8.60) | 3.11 (10.39)
  Social Roles and Activities: number analyzed (Participants) | 45 | 11
  Social Roles and Activities | -1.94 (8.97) | -9.72 (13.05)
  Pain Interference: number analyzed (Participants) | 45 | 11
  Pain Interference | 4.95 (7.17) | 5.91 (8.98)
  Pain Intensity: number analyzed (Participants) | 45 | 11
  Pain Intensity | 1.7 (2.2) | 1.4 (3.6)

10. Secondary Outcome: Mean Change in Health Domains Assessed by PROMIS-29 Scale From Baseline to 24 Months
Description: as for outcome 6
Time Frame: From baseline to 24 months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Subjects Using BurstDR SCS Systems | Subjects Using DRG Systems
Number analyzed (Participants) | 85 | 15
score on a scale
  Physical Function: number analyzed (Participants) | 23 | 7
  Physical Function | -2.75 (7.34) | -4.80 (8.47)
  Anxiety: number analyzed (Participants) | 23 | 7
  Anxiety | 1.99 (11.53) | 3.50 (6.94)
  Depression: number analyzed (Participants) | 23 | 7
  Depression | 0.69 (10.42) | 3.03 (5.28)
  Fatigue: number analyzed (Participants) | 23 | 7
  Fatigue | 2.29 (11.55) | 2.90 (10.83)
  Sleep Disturbance: number analyzed (Participants) | 23 | 7
  Sleep Disturbance | 3.57 (9.53) | 1.31 (8.37)
  Social Roles and Activities: number analyzed (Participants) | 23 | 7
  Social Roles and Activities | -3.09 (11.38) | -3.94 (8.49)
  Pain Interference: number analyzed (Participants) | 23 | 7
  Pain Interference | 7.15 (8.12) | 5.80 (8.22)
  Pain Intensity: number analyzed (Participants) | 23 | 7
  Pain Intensity | 2.0 (2.5) | 2.4 (2.8)

11. Secondary Outcome: Mean Change in Pain Assessed by Pain Catastrophizing Scale (PCS) From Baseline to 3 Months
Description: The PCS is a validated, 13-item scale that evaluates 3 domains of pain-related negative thoughts (rumination, magnification, and helplessness). Subjects rate how often they have the given thought from 0 "not at all" to 4 "all the time". The total score is a sum of all responses, ranging from 0-52. Each domain has a sub-scale score calculated as a sum of the constituent responses with ranges of 0-16 for rumination, 0-12 for magnification, and 0-24 for helplessness.
Time Frame: From baseline to 3 months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Subjects Using BurstDR SCS Systems | Subjects Using DRG Systems
Number analyzed (Participants) | 73 | 15
score on a scale | 15.8 (12.7) | 15.2 (13.3)

12. Secondary Outcome: Mean Change in Pain Assessed by Pain Catastrophizing Scale (PCS) From Baseline to 6 Months
Description: as for outcome 11
Time Frame: From baseline to 6 months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Subjects Using BurstDR SCS Systems | Subjects Using DRG Systems
Number analyzed (Participants) | 67 | 14
score on a scale | 16.1 (12.4) | 14.6 (17.8)

13. Secondary Outcome: Mean Change in Pain Assessed by Pain Catastrophizing Scale (PCS) From Baseline to 12 Months
Description: as for outcome 11
Time Frame: From baseline to 12 months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Subjects Using BurstDR SCS Systems | Subjects Using DRG Systems
Number analyzed (Participants) | 66 | 13
score on a scale | 17.0 (14.6) | 14.0 (17.6)

14. Secondary Outcome: Mean Change in Pain Assessed by Pain Catastrophizing Scale (PCS) From Baseline to 18 Months
Description: as for outcome 11
Time Frame: From baseline to 18 months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Subjects Using BurstDR SCS Systems | Subjects Using DRG Systems
Number analyzed (Participants) | 45 | 11
score on a scale | 14.2 (13.8) | 16.2 (17.7)

15. Secondary Outcome: Mean Change in Pain Assessed by Pain Catastrophizing Scale (PCS) From Baseline to 24 Months
Description: as for outcome 11
Time Frame: From baseline to 24 months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Subjects Using BurstDR SCS Systems | Subjects Using DRG Systems
Number analyzed (Participants) | 23 | 7
score on a scale | 10.7 (11.8) | 19.6 (15.5)

16. Secondary Outcome: Mean Change in Attention to Pain Assessed by Pain Vigilance and Awareness Questionnaire (PVAQ) From Baseline to 3 Months
Description: 'The PVAQ is a validated, 16-item scale that evaluates attention to pain. Subjects rate how frequently each statement represents their experience over the last 2 weeks from 0 "never" to 5 "always". Item scores are summed to produce the total score, which ranges from 0-80 with a higher score indicating greater attention to pain.'
Time Frame: From baseline to 3 months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Subjects Using BurstDR SCS Systems | Subjects Using DRG Systems
Number analyzed (Participants) | 74 | 15
score on a scale | 34.5 (11.9) | 33.1 (13.4)

17. Secondary Outcome: Mean Change in Attention to Pain Assessed by Pain Vigilance and Awareness Questionnaire (PVAQ) From Baseline to 6 Months
Description: as for outcome 16
Time Frame: From baseline to 6 months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Subjects Using BurstDR SCS Systems | Subjects Using DRG Systems
Number analyzed (Participants) | 67 | 14
score on a scale | 35.4 (11.9) | 34.7 (17.6)

18. Secondary Outcome: Mean Change in Attention to Pain Assessed by Pain Vigilance and Awareness Questionnaire (PVAQ) From Baseline to 12 Months
Description: as for outcome 16
Time Frame: From baseline to 12 months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Subjects Using BurstDR SCS Systems | Subjects Using DRG Systems
Number analyzed (Participants) | 66 | 13
score on a scale | 36.0 (12.2) | 33.1 (14.3)

19. Secondary Outcome: Mean Change in Attention to Pain Assessed by Pain Vigilance and Awareness Questionnaire (PVAQ) From Baseline to 18 Months
Description: as for outcome 16
Time Frame: From baseline to 18 months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Subjects Using BurstDR SCS Systems | Subjects Using DRG Systems
Number analyzed (Participants) | 45 | 11
score on a scale | 33.6 (12.3) | 30.5 (15.7)

20. Secondary Outcome: Mean Change in Attention to Pain Assessed by Pain Vigilance and Awareness Questionnaire (PVAQ) From Baseline to 24 Months
Description: as for outcome 16
Time Frame: From baseline to 24 months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Subjects Using BurstDR SCS Systems | Subjects Using DRG Systems
Number analyzed (Participants) | 23 | 7
score on a scale | 32.7 (14.4) | 35.0 (20.4)

21. Secondary Outcome: Change in Pain Condition-related Medication Use From Baseline to 3 Months
Description: Details will be collected regarding dosages and categories of pain-related medication.
Time Frame: From baseline to 3 months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: Morphine milligram equivalent (MME)
Arm/Group | Subjects Using BurstDR SCS Systems | Subjects Using DRG Systems
Number analyzed (Participants) | 44 | 5
Morphine milligram equivalent (MME) | 9.9 (43.4) | 26.4 (59.0)

22. Secondary Outcome: Change in Pain Condition-related Medication Use From Baseline to 6 Months
Description: Details will be collected regarding dosages and categories of pain-related medication.
Time Frame: From baseline to 6 months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: Morphine milligram equivalent (MME)
Arm/Group | Subjects Using BurstDR SCS Systems | Subjects Using DRG Systems
Number analyzed (Participants) | 39 | 5
Morphine milligram equivalent (MME) | 15.6 (51.5) | 33.0 (82.4)

23. Secondary Outcome: Change in Pain Condition-related Medication Use From Baseline to 12 Months
Description: Details will be collected regarding dosages and categories of pain-related medication.
Time Frame: From baseline to 12 months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: Morphine milligram equivalent (MME)
Arm/Group | Subjects Using BurstDR SCS Systems | Subjects Using DRG Systems
Number analyzed (Participants) | 38 | 5
Morphine milligram equivalent (MME) | 16.4 (49.4) | 33.0 (82.4)

24. Secondary Outcome: Change in Pain Condition-related Medication Use From Baseline to 18 Months
Description: Details will be collected regarding dosages and categories of pain-related medication.
Time Frame: From baseline to 18 months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: Morphine milligram equivalent (MME)
Arm/Group | Subjects Using BurstDR SCS Systems | Subjects Using DRG Systems
Number analyzed (Participants) | 85 | 15
Morphine milligram equivalent (MME) | 18.3 (56.6) | 58.9 (84.9)

25. Secondary Outcome: Change in Pain Condition-related Medication Use From Baseline to 24 Months
Description: Details will be collected regarding dosages and categories of pain-related medication.
Time Frame: From baseline to 24 months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: Morphine milligram equivalent (MME)
Arm/Group | Subjects Using BurstDR SCS Systems | Subjects Using DRG Systems
Number analyzed (Participants) | 85 | 15
Morphine milligram equivalent (MME) | 15.4 (31.8) | 90.0 (127.3)

ADVERSE EVENTS:
Time Frame: 2 Year
Arm/Group | Subjects Using BurstDR SCS Systems | Subjects Using DRG Systems
All-Cause Mortality (participants affected / at risk) | 3/85 | 0/15
Serious Adverse Events (participants affected / at risk) | 1/85 | 2/15
Other Adverse Events (participants affected / at risk) | 11/85 | 4/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Subjects Using BurstDR SCS Systems (N=85) | Subjects Using DRG Systems (N=15)
Cerebrospinal Fluid (CSF) Leakage (Nervous system disorders) | 1 | 0
Neuropraxia (Nervous system disorders) | 1 | 0
Pain Below the Level of The Implant (Surgical and medical procedures) | 0 | 1
Weakness, Clumsiness, or Numbness Below the Level of The Implant (Surgical and medical procedures) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Subjects Using BurstDR SCS Systems (N=85) | Subjects Using DRG Systems (N=15)
Battery Failure (Product Issues) | 2 | 0
Persistent Pain at the IPG Site (Injury, poisoning and procedural complications) | 2 | 0
Lead Fracture (General disorders) | 1 | 2
Pain at Anchor Site (Injury, poisoning and procedural complications) | 1 | 0
Post Procedural Pain (Injury, poisoning and procedural complications) | 1 | 0
Sensation of Heat (Product Issues) | 1 | 0
Shocking Sensation (Product Issues) | 1 | 0
Skin Erosion at the IPG Site (Product Issues) | 1 | 0
Thoracic Pain (General disorders) | 1 | 0
Lead Migration, Causing Changes in Stimulation or Reduced Pain Relief (Product Issues) | 2 | 3
Burning in Feet (General disorders) | 0 | 1
High Impedance (Product Issues) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-01-23): https://cdn.clinicaltrials.gov/large-docs/76/NCT03908476/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-03): https://cdn.clinicaltrials.gov/large-docs/76/NCT03908476/SAP_001.pdf